CLINICAL TRIAL: NCT00153725
Title: Intravenous Pantoloc In Aspirin-Induced Ulcer Bleeding
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Chinese University of Hong Kong (Other)
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: PPA Study
Record Dates: First submitted 2005-09-08; First posted 2005-09-12 (Estimated); Last update posted 2006-10-27 (Estimated); Status verified 2006-10

CONDITIONS: Cardiovascular Disease; Cerebrovascular Disorders
MeSH Terms: conditions — Cardiovascular Diseases; Cerebrovascular Disorders | interventions — Aspirin

INTERVENTIONS:
Drug: Aspirin and Pantoloc

SUMMARY:
The aim of the study is to investigate whether intravenous infusion of pantoprazole (Pantoloc) is effective in preventing recurrent bleeding in patients who present with acute ulcer bleeding and continue to use aspirin

DETAILED DESCRIPTION:
Aspirin is an effective treatment for acute stroke and heart attack. However, aspirin also induces ulcer and provokes acute ulcer bleeding. Thus, aspirin is often withheld in acute ulcer bleeding but this precipitate recurrent stroke or heart attack. We previously showed that intravenous infusion of a potent acid suppressant substantially reduced the incidence of recurrent ulcer bleeding in patients who withheld aspirin. The aim of this study is to investigate whether intravenous infusion of an acid suppressant (Pantoprazole) is effective in preventing recurrent ulcer bleeding with continuous use of aspirin.

ELIGIBILITY:
Inclusion Criteria:

* Patients received daily anti-platelet therapy for vascular prophylaxis before admission and will continue need to do so
* Patinets with bleeding peptic ulcers;ulcer actively bleeding or with SRH (Forrest I, IIa and IIb ulcers)
* Endoscopic haemostasis achieved

Exclusion Criteria:

* Presence of ulcer complication precluding endoscopic treatment such as gastric outlet obstruction or ulcer perforation mandating surgical intervention.
* Concomitant use of anticoagulant, NSAIDs or steroid
* Pending to undergo cardiac interventions that need double anti-platelet agent
* Pregnancy
* Terminal illness, or cancer

Ages: 18 Years to 90 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 156
Dates: Start 2003-02; Study Completion 2006-09

PRIMARY OUTCOMES:
Primary Outcome:
Recurrent upper gastrointestinal bleeding within 30 days

CONTACTS AND LOCATIONS:
Overall Officials: Joseph J Sung, MD, Principal Investigator — Chinese University of Hong Kong
Locations (3):
- China (3):
  - Endoscopy Center, North District Hospital, Hong Kong
  - Endoscopy Center, Prince of Wales Hospital, Hong Kong
  - Endoscopy Center, United Christian Hospital, Hong Kong

REFERENCES:
- [Derived] Sung JJ, Lau JY, Ching JY, Wu JC, Lee YT, Chiu PW, Leung VK, Wong VW, Chan FK. Continuation of low-dose aspirin therapy in peptic ulcer bleeding: a randomized trial. Ann Intern Med. 2010 Jan 5;152(1):1-9. doi: 10.7326/0003-4819-152-1-201001050-00179. Epub 2009 Nov 30. PMID 19949136